CLINICAL TRIAL: NCT07389785
Title: Age Related Chromatin Remodelling as a Therapeutic Target for Organ Protection in Cardiac Surgery
Acronym: EPI-CARD
Status: Active, not recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 1086; 356697 (Other: Health Research Authority)
Record Dates: First submitted 2025-09-17; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Surgery; Organ Protection; Ageing
Keywords: chromatin; cardiac surgery; organ protection; multiple long-term conditions; ageing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood, biopsies (right atrial, vascular, adipose tissue and bone marrow).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- MARACAS: Prospective, single-centre observational case-control study.
  Interventions: Other: other
- REDWASH: A multicenter parallel-group randomized controlled trial.
  Interventions: Other: other
- REVAKI-2: Phase IIB placebo-controlled randomised clinical trial.
  Interventions: Other: other
- OB-CARD: Prospective, single-centre case control study.
  Interventions: Other: other
- COPTIC-2: Retrospective, single-centre observational cohort trial.
  Interventions: Other: other
- VAL-CARD: Single-centre, unblinded, randomised controlled trial (Phase 2b).
  Interventions: Other: other
- PRE-OP ENERGY: Single-centre, unblinded, parallel group, randomised controlled trial.
  Interventions: Other: other

INTERVENTIONS:
Other: other — This is not an interventional study.

SUMMARY:
People who have multiple long-term conditions (MLTC) like kidney disease or lung disease are at higher risk of developing organ damage and poor quality of life following heart surgery. Decades of research have failed to identify drugs or treatments that prevent this.

Our research has shown that people with MLTC have changes in their heart cells before surgery that are referred to by researchers as Biological Ageing. These changes combine to make people with MLTC more susceptible to organ damage after heart surgery, have delayed recovery, and lower quality of life.

This research programme will investigate the processes linking MLTC, changes in heart cells, and organ damage.

Our previous research suggests that MLTC lead to the infiltration of white cells from the blood into the heart muscle, a process called inflammageing. This alters the DNA in heart cells, reduces their pumping function and leaves them more likely to be damaged by surgery.

We have also shown that these changes are affected by obesity. We have also shown that changes in other types of heart cells with ageing are associated with damage to the lining of blood vessels, bleeding and damage to the kidneys.

We will use existing clinical data from previous studies and molecular data from heart cells obtained at surgery to better understand the molecular changes underlying our previous observations. This includes data from previous trials of drugs and dietary modification that aimed to modify the cellular DNA changes caused by inflammageing.

Using external data, we will check whether similar results are evident in other studies. We will then select the most likely processes underlying our observations and test whether these relationships are causal using genomic analysis and the UK Biobank data. Finally, we will use established analytical methods to identify potential drugs that may target these processes.

Positive results will provide a better understanding of the heart damage that is often seen in people with MLTC as well as new treatments for evaluation on further research.

DETAILED DESCRIPTION:
Organ injury is common following cardiac surgery, where it contributes to excess mortality, delayed recovery, progression of LTC, poor quality of life, and increased use of healthcare resources.

People with MLTC demonstrate increased susceptibility to organ injury and its complications. Using a multi-omics approach we have shown that MLTC are associated with biological ageing in human myocardium. Using snRNAseq, we have shown that progression of MLTC are associated with acceleration of biological ageing, characterised by T cell exhaustion, dysregulated tissue resident macrophage activation, and increased susceptibility of cardiomyocytes to metabolic stress.

Genetic modification of these processes altered susceptibility to 90-day mortality following cardiac surgery in UK Biobank. Reversal of biological ageing mechanisms including mTOR activation, histone modification, disabled autophagy, or cell senescence reduces the susceptibility of myocardium to ischaemia reperfusion injury in mice. These observations lead us to hypothesise that pre-surgery reversal of biological ageing may have organ protective effects.

Cellular ageing is characterised by changes in chromatin accessibility that are determined by histone DNA interaction. The interaction between histones and DNA in the nucleosome determine the accessibility of promoters, enhancers, and transcription factors to molecular DNA and subsequently gene expression. Reversal of age-related changes in chromatin prevents cardiac ageing in mice.

In preliminary work we have shown that genetic modification underlying biological ageing in human myocardial biopsies is determined in part by changes in chromatin accessibility. We have shown associations between MLTC including obesity, genetic modification, and organ injury affecting the heart, kidney and vascular endothelium (bleeding). We now propose to comprehensively characterise the changes in chromatin accessibility, gene expression, cell secretomes and cell-cell interactions and single cell resolution that underly these observations.

This will be the first study to use integrated multi-omics to identify cellular phenotypes associated with different stages of biological ageing. The study will explore the contribution of a central hallmark of biological ageing; chromatin accessibility. Observational data from multi-omics snRNAseq and snATACseq will be validated in external datasets, and the causal effect of chromatin accessibility of susceptibility to organ injury will be explored using secondary analyses of RCTs. This research represents a first in man analysis of the role of chromatin remodelling in myocardial ageing and susceptibility to organ injury.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing cardiac surgery with cardiopulmonary bypass (CPB) enrolled in seven clinical studies in five UK centres.

Exclusion Criteria:

* Patients who did not consent to participate in the included trials, or participants who did not consent for secondary research of their data and samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cardiac surgery patients.
Sampling Method: Non-Probability Sample
Enrollment: 3055 (Actual)
Dates: Start 2025-09-29 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Study 1 | 5 years
  For the clinical studies, outcomes will be restricted to those measured prospectively in the individual studies.
  For the UK Biobank data, the primary outcome is time to death or emergency re-hospitalisation requiring overnight admission within 365 days following discharge after major surgery.
Study 2 | 5 years
  The analysis will identify differentially expressed genes, gene pathways, and networks in cell types by phenotype. The data will also identify differences in promoter accessibility by cell type and phenotype
Study 3 | 5 years
  These studies will provide quantitative targeted validation of genes, proteins and DNA accessibility by cell type and phenotype in human myocardial biopsies obtained at surgery in the listed studies.
  We will identify anonymised publicly available external data sources that have evaluated biological ageing and inflammageing in human tissues. We will duplicate our primary genomics analysis in this secondary dataset.
Study 4 | 5 years
  We will quantify the effects of genetic modification of key genes and pathways identified in Studies 1-3 on mortality and freedom from hospitalisation in UK Biobank.
Study 5 | 48 hours post-operation
  Clinical outcomes: Area under the troponin curve from baseline to 48 hours post-surgery.
Study 5 | 72 hours post-operation
  Clinical outcomes: Area under the creatinine curve from baseline to 72 hours post-surgery.
Study 5 | 6 weeks
  Process outcomes: Valproate exposure
Study 5 | 6 weeks
  Process outcomes: Calorific intake
Study 5 | 6 weeks
  Process outcomes: Weight gain.
Study 5 | 1 day (operation day)
  Experimental Outcomes: Combined snRNAseq/ ATACseq in myocardial biopsies (5 per group) obtained at surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin J Murphy, BSc, MBChB, FRCS, MD, FRCS CTh, Principal Investigator — University of Leicester
Locations (1):
- University of Leicester, Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided